CLINICAL TRIAL: NCT01583569
Title: Complex Dynamic Systems in Mood Disorders
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director of Research, Bipolar Clinic and Research Program, Massachusetts General Hospital
Other Study IDs: 3273723; 1K18MH093939-01 (NIH)
Record Dates: First submitted 2012-03-30; First posted 2012-04-24 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
Keywords: Complex Dynamic Systems; Biomarkers; Mood Disorders
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Mood Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Complex Dynamic Systems in Mood Disorders is an observational, exploratory study of the relationship between voice samples, heart rate, respiration, movement, galvanic skin conductance, and sleep architecture with mood states in patients with Major Depressive Disorder, Bipolar Disorder, and healthy controls. The overall hypothesis is that nonlinear dynamic analyses will be able to reveal hidden patterns of complexity in each domain of voice, heart rate variability, movement, arousal, and sleep stage data.

DETAILED DESCRIPTION:
Aim 1: To assess multichannel physiologic measures associated with mood disorders.

Hypothesis: The overall hypothesis is that nonlinear dynamic analyses will be able to reveal hidden patterns of complexity in each domain of voice, heart rate variability (RR intervals), movement, arousal, and sleep stage data.

Aim 2: To assess differences in patterns and complexity of multiple physiological measures in patients with MDD compared to healthy controls.

Hypothesis: MDD will be associated with decreased measures of complexity and increased measures of approximate entropy compared to healthy controls.

Aim 3: To assess differences in patterns and complexity of multiple physiologic measures in patients with BD compared to healthy controls.

Hypothesis: BD will be associated with decreased measures of complexity and increased measures of approximate entropy compared to healthy controls.

Aim 4: To assess changes in patterns and complexity of multiple physiologic measures at baseline and after 2 weeks of treatment for patients with MDD and BD.

Hypothesis: Measures of complexity will increase and measures of approximate entropy will decrease in the first two weeks of treatment.

Aim 5: To assess the relationship between changes in patterns and complexity of multiple physiologic measures and changes in mood state.

Hypothesis: Measures of complexity will increase and measures of approximate entropy will decrease, especially for those who are much or very much improved

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 65.
* Meet DSM-IV criteria for MDD (n=5), BD (n=5), or healthy controls with no psychiatric diagnosis (n=5).
* Willing and able to wear a wearable device to measure sleep parameters
* Willing and able to provide voice samples.
* Subjects with MDD must not be taking psychiatric medications at the time of evaluation.Subjects with BD can be taking psychiatric medications, since it is not feasible for patients with BD to be completely free of mood stabilizing medications. These medications will be limited to lithium, second generation antipsychotics.
* Currently a patient or research participant at the DCRP or the BCRP or are healthy controls enrolled in evaluation studies.

Exclusion Criteria:

* Primary sleep disorder, including restless legs syndrome, difficulties in initiating and maintaining sleep.
* Movement disorders (e.g. Parkinson's, Huntington's, tardive dyskinesia, primary chorea).
* Active substance abuse or dependence in the past 3 months.
* Cardiovascular or pulmonary disease, including uncontrolled hypertension, arrhythmias, history of myocardial infarction, asthma, COPD, or pulmonary carcinoma.
* Cardiovascular or pulmonary medications (aspirin and statins are allowable).
* Anticonvulsants.
* Sedative/hypnotics (e.g. benzodiazepines, eczopiclone).
* Smokers.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will consist of subjects with Major Depressive Disorder(n=5), Bipolar Disorder (n=5), as well as healthy controls (n=5)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bipolar Clinic and Research Program at Massachusetts General Hospital, Boston, Massachusetts, United States